CLINICAL TRIAL: NCT07363824
Title: A Study on the Correlation Between Tear Iron Levels and the Severity of Dry Eye Disease.
Status: Recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Ruili Wei, Chief of Ophthalmology, Shanghai Changzheng Hospital
Other Study IDs: DED-A
Record Dates: First submitted 2026-01-05; First posted 2026-01-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease; Iron
Keywords: DED; iron
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CON
  Interventions: Procedure: Diagnostic tear fluid collection and ocular surface evaluation
- DED
  Interventions: Procedure: Diagnostic tear fluid collection and ocular surface evaluation

INTERVENTIONS:
Procedure: Diagnostic tear fluid collection and ocular surface evaluation — This is an observational study; no therapeutic intervention is administered. All participants undergo a single, standardized study visit that includes:
  Tear Fluid Collection: Tear samples are collected using sterile Schirmer test strips (without anesthesia) placed in the lower conjunctival sac for 5 minutes.
  Comprehensive Ocular Surface Evaluation:
  Symptom Assessment: Completion of the Ocular Surface Disease Index (OSDI) questionnaire.
  Clinical Tests: Measurement of fluorescein tear film breakup time (FBUT), corneal fluorescein staining (CFS) scoring, and Schirmer I test.
  The collected tear samples are subsequently analyzed for iron concentration. All procedures are diagnostic and evaluative in nature.

SUMMARY:
This study aims to see if the amount of iron in tears is linked to how severe dry eye disease is. We hope this can lead to a new way to help diagnose and understand dry eye. This is an observational study. We will compare tear samples from people with dry eye to samples from people with healthy eyes. We will measure the iron content in the tears and see if it correlates with standard dry eye test results and symptom scores.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years, inclusive.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* History or clinical suspicion of significant systemic conditions: hematologic diseases, severe systemic infections, malignancies (treated or untreated), or chronic hepatic/renal insufficiency.
* Use of artificial tears or any topical eye drops within 2 hours prior to examination.
* Active ocular allergy, infection, or severe blepharitis within the past 1 month.
* Systemic or topical use of antibiotics, corticosteroids, NSAIDs, or immunosuppressants within the past 1 month.
* History of contact lens wear within the past 1 month.
* History of blood transfusion, ocular surgery, or significant ocular trauma within the past 6 months.
* Women who are pregnant, breastfeeding, or postmenopausal women undergoing hormone replacement therapy.
* Known hypersensitivity to fluorescein sodium.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Based on your study protocol, here is the description for the "Study Population Description" field:
  This single-center, cross-sectional study will recruit participants from the patient population and staff/community at the Ophthalmology Department of Shanghai Changzheng Hospital. The Dry Eye Disease (DED) group will consist of consecutive patients presenting to the clinic who are diagnosed with DED according to the 2024 Chinese Expert Consensus criteria. The healthy control group will be recruited through hospital staff volunteers and community advertisements. All participants will be enrolled during the specified study period from the single site.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between tear fluid iron concentration and dry eye symptom severity | baseline
  The strength of association between the concentration of iron (in μg/mL) in tear fluid collected via Schirmer strips and the total score on the Ocular Surface Disease Index (OSDI) questionnaire.

SECONDARY OUTCOMES:
Correlation between tear fluid iron concentration and tear film stability | baseline
  The correlation between tear iron concentration and fluorescein tear film breakup time (FBUT) measured in seconds.
Correlation between tear fluid iron concentration and tear secretion volume | baseline
  The correlation between tear iron concentration and the result of the Schirmer I test (without anesthesia) measured in millimeters of wetting over 5 minutes.
Correlation between tear fluid iron concentration and corneal epithelial damage | baseline
  The correlation between tear iron concentration and the Corneal Fluorescein Staining (CFS) score, a standardized clinical grading of epithelial damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No